CLINICAL TRIAL: NCT03927365
Title: Muco-ciliary Cleansing of Lungs in COPD With and Without a Salt Particle Inhaler
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Liita Care ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LC.001
Record Dates: First submitted 2018-10-01; First posted 2019-04-25 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: COPD; Copd Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants cross over from active to placebo or vice versa in random order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization of a salt particle inhaler devices with (active) or without (placebo) content
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt particle inhaler with content (Active Comparator): Participants inhaling from a salt particle inhaler with content
  Interventions: Device: Inhalation from a salt particle inhaler with or without content
- Salt particle inhaler without content (Placebo Comparator): Participants inhaling from a salt particle inhaler without content
  Interventions: Device: Inhalation from a salt particle inhaler with or without content

INTERVENTIONS:
Device: Inhalation from a salt particle inhaler with or without content — Inhalation from inhaler with (active) or without (placebo) content

SUMMARY:
Cross-over trial of the effect of a salt particle inhaler on pulmonary muco-ciliary cleansing in COPD patients as measured by lung scintigraphy.

DETAILED DESCRIPTION:
Stable COPD patients will be examined twice with minimum two, maximum 14 days interval. In randomized order the patients will inhale from a salt particle inhaler with (active) or without (placebo) content.

ELIGIBILITY:
Inclusion Criteria:

* COPD grade 1, 2 and 3 in stable condition (less than 10% change of FEV1 ratio between investigation visits

Exclusion Criteria:

* Pregnant or lactating women
* Patients exposed to radionuclear isotopes within one month
* Patients under antibiotic treatment
* Patients with known hyper reactive airways

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Muco-ciliary clearance | Activity at time zero
  Retention of inhaled radioactive marker in percentage
Muco-ciliary clearance | Activity at time 30 minutes
  Retention of inhaled radioactive marker in percentage
Muco-ciliary clearance | Activity at time 90 minutes
  Retention of inhaled radioactive marker in percentage
Muco-ciliary clearance | Activity at time 120 minutes
  Retention of inhaled radioactive marker in percentage

SECONDARY OUTCOMES:
Registering number of coughs | Activity at any time between time zero and 120 minutes
  Number of coughs during investigation is noted
Collection of sputum | Activity at any time between time zero and 120 minutes
  Sputum during investigation is collected for analysis of radioactivity content
Symptoms in the subjects health | Activity at time zero
  Subjective symptom description during last 24 hours is done by a CCQ (Clinical COPD Questionnaire)
Symptoms in the subjects health | Activity at time 30
  Subjective symptom description during investigation is done by a questionnaire
Symptoms in the subjects health | Activity at time 120
  Subjective symptom description during investigation is done by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jann Mortensen, MD Professor, Principal Investigator — Rigshospitalet, Clin Nuclear & Physiolog dept.
Locations (1):
- Rigshospitalet, Clin nuclear and physiolog dept., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No